CLINICAL TRIAL: NCT06296888
Title: Radiofrequency Balloon Catheter Ablation for Atrial Fibrillation: Durability of Pulmonary Vein Isolation and Clinical Outcome - The RABAAF Study
Brief Title: Radiofrequency Balloon Ablation for Atrial Fibrillation: Durability of Pulmonary Vein Isolated and Clinical Outome
Acronym: RABAAF
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jim Hansen (Other)
Collaborators: University Hospital, Gentofte, Copenhagen (Other); Biosense Webster, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Jim Hansen, Consultant Cardiologist, MD, DMSc, University Hospital, Gentofte, Copenhagen
Organization: University Hospital, Gentofte, Copenhagen (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P-2022-673; 2203718 (Other: De Videnskabsetiske Medicinske Komiteer)
Record Dates: First submitted 2024-02-28; First posted 2024-03-06 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-02

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Radiofrequency balloon catheter ablation (Experimental): Enrolled patients will undergo PVI by radiofrequency balloon ablation.
  Interventions: Procedure: Radiofrequency balloon catheter ablation

INTERVENTIONS:
Procedure: Radiofrequency balloon catheter ablation — Radiofrequency balloon ablation using the HELIOSTAR™ ablation catheter.

SUMMARY:
Atrial fibrillation (AF) is the most common heart rhythm disorder affecting 2-4% of the adult human population. AF is a disturbance in the electrical impulses of the heart - an electrical disturbance commonly originating from the pulmonary veins.

Normalization of the heart rhythm with anti-arrhythmic drugs often fail and is frequently associated with side effects. Therefore, a treatment termed ablation by catheters via an inguinal vein has been devised and is increasingly being used for the treatment of AF. The cornerstone of this treatment is electrical isolation of the pulmonary veins so that the nocuous electrical impulses from the pulmonary veins cannot cause a disturbance in the heart rhythm and initiate episodes of AF. This treatment is called pulmonary vein isolation (PVI). Recent studies have shown that PVI is better than anti-arrhythmic drug treatment in the prevention of recurrence of AF, but despite substantial improvements in techniques and tools only 60-70% are cured from AF by a single PVI procedure, and in around 80% of patients who require additional catheter ablation, durable isolation of all the pulmonary veins has not been achieved. Improved tools for durable PVI are therefore required.

A novel catheter to achieve PVI called the HELIOSTAR™ radiofrequency balloon ablation catheter has shown promising clinical results with a favorable safety profile, but the durability of PVI has not been evaluated. Therefore, we aim to investigate the long-term durability of PVI by the radiofrequency balloon and the clinical outcome following the procedure.

In this study, patients with AF referred for catheter ablation will undergo an initial PVI treatment using the radiofrequency balloon catheter. All patients will undergo a repeat electrophysiology (EP) study after 4-6 months to determine to durability of PVI. Patients will be issued with a 48-hour heart rhythm monitor at 3 and 12 months after the initial PVI. Patients-reported effects on quality of life by AF related symptoms will be evaluated using a specialized questionnaire provided approximately every third month throughout the 12 month follow-up.

DETAILED DESCRIPTION:
The study is a single-arm prospective cohort study in 45 patients referred for AF ablation that will assess the durability of PVI, freedom from atrial tachyarrhythmia (ATA) recurrence and patient reported quality of life following PVI by radiofrequency balloon catheter ablation.

All patients, irrespective of ATA recurrence, will undergo a repeat EP study 4-6 months after initial PVI for the assessment of PVI durability. Recurrence of ATA after the initial PVI will be evaluated by 48-hour ambulatory electrocardiography (ECG) monitoring following a 3-months blanking period after the PVI procedure, and effect on quality of life will be evaluated by questionnaires at baseline, 3 months after the initial PVI, and at the time of the repeat procedure.

Recurrence of ATA after the repeat EP study will be evaluated by 48-hour ambulatory ECG monitoring 12 months after the initial PVI, and effect on quality of life will be evaluated by additional questionnaires at 9 and 12 months after the initial PVI.

In patients with symptoms of potentiel ATA outside the protocolled ambulatory ECG monitoring periods, ECG diagnostics appropriate for the duration and frequency of episodes with symptoms will be utilized.

ELIGIBILITY:
Inclusion Criteria:

* Documented AF
* Clinical indication for ablation
* First time AF ablation
* Scheduled for PVI only

Exclusion Criteria:

* Contraindication for ablation
* Inability to give informed consent
* Documented atrial flutter or any other arrhythmia requiring ablation in addition to PVI
* Known esophageal or nasopharyngeal pathology that would preclude insertion of an esophageal temperature probe
* Severe asthma that would preclude adenosine injections for assessment of dormant conduction

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-03-15 (Estimated); Study Completion 2024-08-09 (Estimated)

PRIMARY OUTCOMES:
Proportion of durably isolated PVs observed at repeat EP study | 4-6 months
  During repeat EP study 4-6 months after initial PVI, all PVs are assessed for bidirectional block. Any reconnected PVs will be reisolated. After confirmation of bidirectional conduction block (preceded by reisolation in case of PV reconduction), adenosine injections will be used to test for dormant conduction. PVs with dormant conduction are not considered durably isolated.

SECONDARY OUTCOMES:
Proportion of patients with durable isolation of all PVs observed at repeat EP study | 4-6 months
  During repeat EP study 4-6 months after initial PVI, all PVs are assessed for bidirectional block. Any reconnected PVs will be reisolated. After confirmation of bidirectional conduction block (preceded by reisolation in case of PV reconduction), adenosine injections will be used to test for dormant conduction. PVs with dormant conduction are not considered durably isolated.
Proportion of patients remaining free from recurrence of ATA after the initial PVI | 4-6 months
  The proportion of patients that remain free from recurrence ATA (AF, atrial flutter, and/or atrial tachycardia) ≥ 30 seconds of duration following a 3 month blanking period after initial PVI, documented by any type of ECG.
Difference in the effect of AF related symptoms on quality of life between baseline and after the initial PVI | 4-6 months
  The effect of AF related symptoms on quality of life assessed by the sum of units on The Atrial Fibrillation Effect on QualiTy of life survey (AFEQT) questionnaire
Complications | Occurring within 3 months after the initial PVI procedure
  Complications attributed to radiofrequency balloon catheter ablation

OTHER OUTCOMES:
Proportion of patients remaining free from recurrence of ATA after the repeat EP study | 12 months
  The proportion of patients that remain free from recurrence ATA ≥ 30 seconds of duration following a 3 month blanking period after the repeat EP study, documented by any type of ECG.
Difference in the effect of AF related symptoms on quality of life between baseline, after the initial PVI, and after the repeat EP study | 12 months
  The effect of AF related symptoms on quality of life assessed by the sum of units on AFEQT questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Jim Hansen, MD, DMSc, Principal Investigator — University Hospital, Gentofte, Copenhagen
Locations (1):
- Gentofte Hospital, Hellerup, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hindricks G, Potpara T, Dagres N, Arbelo E, Bax JJ, Blomstrom-Lundqvist C, Boriani G, Castella M, Dan GA, Dilaveris PE, Fauchier L, Filippatos G, Kalman JM, La Meir M, Lane DA, Lebeau JP, Lettino M, Lip GYH, Pinto FJ, Thomas GN, Valgimigli M, Van Gelder IC, Van Putte BP, Watkins CL; ESC Scientific Document Group. 2020 ESC Guidelines for the diagnosis and management of atrial fibrillation developed in collaboration with the European Association for Cardio-Thoracic Surgery (EACTS): The Task Force for the diagnosis and management of atrial fibrillation of the European Society of Cardiology (ESC) Developed with the special contribution of the European Heart Rhythm Association (EHRA) of the ESC. Eur Heart J. 2021 Feb 1;42(5):373-498. doi: 10.1093/eurheartj/ehaa612. No abstract available. PMID 32860505
- [Background] Calkins H, Hindricks G, Cappato R, Kim YH, Saad EB, Aguinaga L, Akar JG, Badhwar V, Brugada J, Camm J, Chen PS, Chen SA, Chung MK, Nielsen JC, Curtis AB, Davies DW, Day JD, d'Avila A, de Groot NMSN, Di Biase L, Duytschaever M, Edgerton JR, Ellenbogen KA, Ellinor PT, Ernst S, Fenelon G, Gerstenfeld EP, Haines DE, Haissaguerre M, Helm RH, Hylek E, Jackman WM, Jalife J, Kalman JM, Kautzner J, Kottkamp H, Kuck KH, Kumagai K, Lee R, Lewalter T, Lindsay BD, Macle L, Mansour M, Marchlinski FE, Michaud GF, Nakagawa H, Natale A, Nattel S, Okumura K, Packer D, Pokushalov E, Reynolds MR, Sanders P, Scanavacca M, Schilling R, Tondo C, Tsao HM, Verma A, Wilber DJ, Yamane T. 2017 HRS/EHRA/ECAS/APHRS/SOLAECE expert consensus statement on catheter and surgical ablation of atrial fibrillation. Heart Rhythm. 2017 Oct;14(10):e275-e444. doi: 10.1016/j.hrthm.2017.05.012. Epub 2017 May 12. No abstract available. PMID 28506916
- [Background] Andrade JG, Wells GA, Deyell MW, Bennett M, Essebag V, Champagne J, Roux JF, Yung D, Skanes A, Khaykin Y, Morillo C, Jolly U, Novak P, Lockwood E, Amit G, Angaran P, Sapp J, Wardell S, Lauck S, Macle L, Verma A; EARLY-AF Investigators. Cryoablation or Drug Therapy for Initial Treatment of Atrial Fibrillation. N Engl J Med. 2021 Jan 28;384(4):305-315. doi: 10.1056/NEJMoa2029980. Epub 2020 Nov 16. PMID 33197159
- [Background] Kuniss M, Pavlovic N, Velagic V, Hermida JS, Healey S, Arena G, Badenco N, Meyer C, Chen J, Iacopino S, Anselme F, Packer DL, Pitschner HF, Asmundis C, Willems S, Di Piazza F, Becker D, Chierchia GB; Cryo-FIRST Investigators. Cryoballoon ablation vs. antiarrhythmic drugs: first-line therapy for patients with paroxysmal atrial fibrillation. Europace. 2021 Jul 18;23(7):1033-1041. doi: 10.1093/europace/euab029. PMID 33728429
- [Background] Wazni OM, Dandamudi G, Sood N, Hoyt R, Tyler J, Durrani S, Niebauer M, Makati K, Halperin B, Gauri A, Morales G, Shao M, Cerkvenik J, Kaplon RE, Nissen SE; STOP AF First Trial Investigators. Cryoballoon Ablation as Initial Therapy for Atrial Fibrillation. N Engl J Med. 2021 Jan 28;384(4):316-324. doi: 10.1056/NEJMoa2029554. Epub 2020 Nov 16. PMID 33197158
- [Background] Reddy VY, Schilling R, Grimaldi M, Horton R, Natale A, Riva S, Tondo C, Kuck KH, Neuzil P, McInnis K, Bishara M, Zhang B, Govari A, Abdelaal A, Mansour M. Pulmonary Vein Isolation With a Novel Multielectrode Radiofrequency Balloon Catheter That Allows Directionally Tailored Energy Delivery: Short-Term Outcomes From a Multicenter First-in-Human Study (RADIANCE). Circ Arrhythm Electrophysiol. 2019 Dec;12(12):e007541. doi: 10.1161/CIRCEP.119.007541. Epub 2019 Dec 12. PMID 31826648
- [Background] Dhillon GS, Honarbakhsh S, Di Monaco A, Coling AE, Lenka K, Pizzamiglio F, Hunter RJ, Horton R, Mansour M, Natale A, Reddy V, Grimaldi M, Neuzil P, Tondo C, Schilling RJ. Use of a multi-electrode radiofrequency balloon catheter to achieve pulmonary vein isolation in patients with paroxysmal atrial fibrillation: 12-Month outcomes of the RADIANCE study. J Cardiovasc Electrophysiol. 2020 Jun;31(6):1259-1269. doi: 10.1111/jce.14476. Epub 2020 Apr 23. PMID 32250514
- [Background] Schilling R, Dhillon GS, Tondo C, Riva S, Grimaldi M, Quadrini F, Neuzil P, Chierchia GB, de Asmundis C, Abdelaal A, Vanderlinden L, Tan T, Ding WY, Gupta D, Reddy VY. Safety, effectiveness, and quality of life following pulmonary vein isolation with a multi-electrode radiofrequency balloon catheter in paroxysmal atrial fibrillation: 1-year outcomes from SHINE. Europace. 2021 Jun 7;23(6):851-860. doi: 10.1093/europace/euaa382. PMID 33450010
- [Background] Sorensen SK, Johannessen A, Worck R, Hansen ML, Hansen J. Radiofrequency Versus Cryoballoon Catheter Ablation for Paroxysmal Atrial Fibrillation: Durability of Pulmonary Vein Isolation and Effect on Atrial Fibrillation Burden: The RACE-AF Randomized Controlled Trial. Circ Arrhythm Electrophysiol. 2021 May;14(5):e009573. doi: 10.1161/CIRCEP.120.009573. Epub 2021 Apr 9. PMID 33835823
- [Background] Worck R, Sorensen SK, Johannessen A, Ruwald M, Haugdal M, Hansen J. Posterior wall isolation in persistent atrial fibrillation feasibility, safety, durability, and efficacy. J Cardiovasc Electrophysiol. 2022 Aug;33(8):1667-1674. doi: 10.1111/jce.15556. Epub 2022 May 31. PMID 35598313
- [Derived] Sorensen SK, Riis-Vestergaard LD, Tonnesen J, Johannessen A, Worck R, Eskesen K, Bertolo G, Mayorga M, Haugdal MA, Ruwald MH, Hansen ML, Hansen J. Durability of Pulmonary Vein Isolation With the Heliostar Radiofrequency Balloon-The Prospective RABAAF Study With Protocol-Mandated Repeat Electrophysiology Studies. J Cardiovasc Electrophysiol. 2025 Sep;36(9):2320-2329. doi: 10.1111/jce.70010. Epub 2025 Jul 15. PMID 40662466